CLINICAL TRIAL: NCT04493996
Title: Increasing Preoperative Cognitive Reserve to Prevent Postoperative Delirium and Postoperative Cognitive Decline in Cardiac Surgical Patients. A Randomized Controlled Trial on Cognitive Training
Brief Title: Increasing Preoperative Cognitive Reserve to Prevent Postoperative Cognitive Dysfunction in Cardiac Surgical Patients
Acronym: INCORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Brain Research Group, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 48/20
Record Dates: First submitted 2020-07-21; First posted 2020-07-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Cognitive Decline; Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: Cardiac Surgery; Postoperative Cognitive Decline; Postoperative Delirium; Cognitive Training; Cognitive Reserve; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training group (Experimental)
  Interventions: Behavioral: Cognitive training
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive training — The cognitive training involves a standardized, paper-and-pencil-based cognitive training that will be performed by the patients at home for approximately 40 minutes per day over a preoperative period of 2-3 weeks
  Arms: Cognitive training group

SUMMARY:
Postoperative delirium (POD) and postoperative cognitive decline (POCD) can be observed after cardiosurgical interventions. Taken together, these postoperative neurocognitive dysfunctions contribute to increased morbidity and mortality and higher economic costs. Preoperative risk factors of postoperative neurocognitive dysfunctions, such as decreased neuropsychometric performance or decreased cognitive daily activities, can be interpreted as reduced cognitive reserve. The aim of this study is to build up cognitive reserves to protect against the development of POD and POCD through preoperative, home-based, cognitive training.

DETAILED DESCRIPTION:
The planned research project is a monocentric, 2-arm randomized controlled intervention study involving 100 patients undergoing elective cardiac surgery with extracorporeal circulation. Patients will be assigned to a training group or control group. The intervention involves a standardized, paper-and-pencil-based cognitive training that will be performed by the patients at home for approximately 40 minutes per day over a preoperative period of 2-3 weeks. The control group will receive neither cognitive training nor a placebo intervention. A detailed assessment of psychological functions will be performed approximately 2-3 weeks before the start of training, at the end of the training, during hospitalization, at discharge from the acute clinic, and 3 months after surgery. The primary objective of this study is to investigate the interventional effect of preoperative cognitive training on the incidence of POD during the stay in the acute clinic, the incidence of POCD at the time of discharge from the acute clinic, and 3 months after surgery. Secondary objectives are to determine the training effect on objective cognitive functions before the surgery and subjective cognitive functions, as well as health-related quality of life 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery (coronary artery bypass surgery, aortic or mitral valve replacement/reconstruction, or combination surgery) with standardized extracorporeal circulation
* A sufficiently good knowledge of German is necessary as cognitive training and neuropsychological tests are language-dependent

Exclusion Criteria:

* History of stroke and preexisting psychiatric or neurological disorders that may impair the neuropsychological performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative cognitive decline at 3 months after surgery, defined as a decrease between pre- and postoperative examinations of one standard deviation in at least 20% of all objective neuropsychological parameters | Immediately pre-training to 3 month post-surgery
  The objective neuropsychological parameters measure cognitive domains like Immediate memory span, free recall, recognition memory, selective attention, working memory, inhibition and word fluency. These cognitive domains will be measured with the following instruments: "Verbaler Lern- und Merkfähigkeitstest" (VLMT), "Brief Visuospatial Memory Test-Revised" (BVMT-R), "Trail Making Test A/B" (TMT), "Letter Number Span Test" (LNS), "Regensburger Wortflüssigkeits-Test" (RWT), and "Syndrom-Kurz Test" (SKT-7).
Number of participants with postoperative cognitive decline at the time of discharge from the acute clinic, defined as a decrease between the pre- and postoperative examinations of one standard deviation measured with the "Montreal Cognitive Assessment" | Immediately pre-training to approximately 1 week post-surgery
  The "Montreal Cognitive Assessment" (MOCA) is a screening procedure for general cognitive function.
Number of participants with postoperative delirium during the stay in the intensive care unit as assessed using the "Intensive Care Delirium Screening Checklist" (ICDSC) | Immediately post-surgery to approximately 1-2 days post-surgery
  Postoperative delirium is defined as the occurrence of at least one delirious episode during a stay in the intensive care unit. The "Intensive Care Delirium Screening Checklist" (ICDSC) record the clinical symptoms of consciousness, attention, orientation, hallucinations, psychomotor retardation or agitation, speech, and changing symptoms by observing behavior and asking concrete questions to the patient.
Number of participants with postoperative delirium during the stay on normal ward as assessed using the "Confusion Assessment Method" (3D-CAM) | Approximately 1 week (Immediately post-intensive care unit to approximately 1 week post-intensive care unit)
  Postoperative delirium is defined as the occurrence of at least one delirious episode during a stay in an intensive care unit or normal ward. The "Confusion Assessment Method" (3D-CAM) record the clinical symptoms of consciousness, attention, orientation, hallucinations, psychomotor retardation or agitation, speech, and changing symptoms by observing behavior and asking concrete questions to the patient.

SECONDARY OUTCOMES:
Change from baseline cognitive failures in everyday life at 3 months after surgery as assessed using the "Cognitive Failures Questionnaire" (CFQ) | Immediately pre-training to 3 month post-surgery
  The "Cognitive Failures Questionnaire" (CFQ) measure the frequency of failures in daily living in terms of memory, attention, action, and perception.
Change from baseline health-related quality of life at 3 months after surgery as assessed using the "36-Item Short Form Health Survey" (SF36) | Immediately pre-training to 3 month post-surgery
  The "36-Item Short Form Health Survey" (SF36) includes 36 questions covering 8 health-related factors: vitality, physical functioning, bodily pain, general health perception, physical role function, emotional role function, social role functioning, and mental health.
Change from baseline visual immediate memory span at the end of cognitive training as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline visual free recall at the end of cognitive training as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline visual recognition memory at the end of cognitive training as assessed using the "Brief Visuospatial Memory Test-Revised" (BVMT-R) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Brief Visuospatial Memory Test-Revised" (BVMT-R), the patient is shown six geometric figures for 10 seconds on a DIN A4 sheet of paper, which are to be drawn directly afterward. This procedure is repeated with the same figures in a total of three learning trials. The figures are to be freely replicated in a time-delayed episode with following recognition help.
Change from baseline verbal immediate memory span at the end of cognitive training as assessed using the "Verbaler Lern- und Merkfähigkeitstest" (VLMT) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Verbaler Lern- und Merkfähigkeitstest" (VLMT), a list of words is learned over five learning trials, which, after a interference word list, is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline verbal free recall at the end of cognitive training as assessed using the "Verbaler Lern- und Merkfähigkeitstest" (VLMT) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Verbaler Lern- und Merkfähigkeitstest" (VLMT), a list of words is learned over five learning trials, which, after a interference word list, is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline verbal recognition memory at the end of cognitive training as assessed using the "Verbaler Lern- und Merkfähigkeitstest" (VLMT) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Verbaler Lern- und Merkfähigkeitstest" (VLMT), a list of words is learned over five learning trials, which, after a interference word list, is to be remembered directly and with a delay of about 20 minutes. With subsequent recognition help, the verbal discrimination ability is measured.
Change from baseline selective attention at the end of cognitive training as assessed using the "Trail Making Test A" (TMT) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Trail Making Test A" (TMT-A), the patient has to connect numbers in ascending order on a test sheet as fast as possible.
Change from baseline verbal working memory at the end of cognitive training as assessed using the "Letter Number Span Test" (LNS) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Letter Number Span Test" (LNS), the patient is supposed to rearrange a mixed sequence of letters and numbers through mental reorganization in such a way that first all numbers and then all letters are to be named in ascending order.
Change from baseline cognitive flexibility at the end of cognitive training as assessed using the "Trail Making Test B" (TMT) | Immediately pre-training to approximately 2-3 weeks post-training
  With the "Trail Making Test B" (TMT-B), the patient's task is to connect numbers and letters alternately in ascending order.
Change from baseline inhibition at the end of cognitive training as assessed using the "Syndrom-Kurz Test" (SKT-7) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Syndrom-Kurz Test" (SKT-7), the patient has to rename a series of letters (e.g., "A" instead of "B," and vice versa).
Change from baseline word fluency at the end of cognitive training as assessed using the "Regensburger Wortflüssigkeits-Test" (RWT) | Immediately pre-training to approximately 2-3 weeks post-training
  In the "Regensburger Wortflüssigkeits-Test" (RWT), the patient has to name in one minute as many words as possible from a certain category.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Butz, Dipl.-Psych., Principal Investigator — Department of Cardiac Surgery, Kerckhoff Clinic Bad Nauheim; Martin Jünemann, Dr.med,M.Sc., Principal Investigator — Clinic for Neurology, University Hospital Gießen; Tibo Gerriets, Prof.Dr.med., Principal Investigator — Department of Neurology, Gesundheitszentrum Wetterau; Markus Schönburg, Prof.Dr.med., Principal Investigator — Department of Cardiac Surgery, Kerckhoff Clinic Bad Nauheim
Locations (1):
- Department of Cardiac Surgery, Kerckhoff-Klinik GmbH, Bad Nauheim, Germany